CLINICAL TRIAL: NCT06971198
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of HSK39004 Dry Powder Inhalation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HSK39004-T1-101
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK39004 (Experimental)
  Interventions: Drug: HSK39004
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK39004 — 0.75~4mg
  Arms: HSK39004
Drug: Placebo — 0.75~4mg
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetic characteristics of HSK39004 dry powder inhalation in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form, understand the trialprocedures, and be willing to comply with all trial procedures andrestrictions;
2. 18 years to 45 years (inclusive), male and female;
3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-26 kg/m2 (inclusive) ;
4. Normal lung function during the screening period, no airway obstruction, FEV1 and forced vital capacity(FVC) are at least 80% of the predicted values;
5. Never smoked or have quit smoking for ≥ 12 months and have a previous smoking history of < 5 pack per years;
6. Subjects are willing to voluntarily use effectivecontraceptives from screening to at least 3 months after the last dose administration.

Exclusion Criteria:

1. Have a history of severe and uncontrolled diseases, such ascardiovascular, respiratory, liver, gastrointestinal, endocrine,hematologic, mental/nervous systems diseases within 3 months prior to screening;
2. Have a history of any malignant tumors;
3. Normal or abnormal vital signs, physical examination, laboratory examination, electrocardiogram, and imageological examination have no clinical significance;
4. Previous or current gastrointestinal, liver, kidney, or other disease known to interfere with drug absorption, distribution, metabolism, or excretion;
5. Acute respiratory infections occurred within 6 weeks before screening and/or before randomization;
6. Have a history of high consumption of grapefruit juice, methylxanthinerich food or beverage within 48 hours before the administration;
7. Average alcohol intake is more than 14 unit per week (1unit=10g alcohol , 1 unit=285 mL 4.9% alcohol beer, or 30 mL 40% alcohol spirit, or 100mL 12% alcohol wine) within the 3 months prior to screening;
8. Have a history of drug abuse prior to screening, or positive urine drug screen at screening;
9. Blood donation (or blood loss) ≥400 mL within 3 months prior to the screening;
10. Subjects who have a allergic to any component of HSK39004 or allergic history;
11. Subjects who use any live vaccine within 30 days prior to screening;
12. Have participated in any clinical investigator within 3 months prior to screening;
13. A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial;
14. Not suitable for this study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
adverse events | From the enrollment of the subjects to 72 hours after the last administration

SECONDARY OUTCOMES:
AUC | from 0 to 72 hours after administration
  area under the concentration-time curve
Cmax | from 0 to 72 hours after administration
  maximum plasma concentration
t1/2 | from 0 to 72 hours after administration
  half-life
Vz/F | from 0 to 72 hours after administration
  apparent volume of distribution
CL/F | from 0 to 72 hours after administration
  apparent clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No